CLINICAL TRIAL: NCT04872634
Title: A Phase I/IIa, Open, Single-Center Clinical Trial Evaluating the Safety and Anti-Tumor Activity of SNK01 (Natural Killer Cells) Administered in Combination With Gemcitabine/Carboplatin or Gemcitabine/Carboplatin/Cetuximab to Locally Advanced or Metastatic Non-small Cell Lung Cancer Patients Who Have Failed Prior Tyrosine Kinase Inhibitor (TKI) Therapy (SNK_ASTER)
Brief Title: A Study to Evaluate the Safety and Anti-tumor Activity of SNK01 (NK Cells) Administered in Combination With Chemotherapy or Chemotherapy / Cetuximab in Local Advanced or Metastatic Non-small Cell Lung Cancer Patients Who Failed Tyrosine Kinase Inhibitor Treatment
Acronym: SNK_ASTER
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NKMAX Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNK01_TRN12a
Record Dates: First submitted 2021-04-21; First posted 2021-05-04 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cytotoxins; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SNK01 (4ⅹ10^9 cells) + GC (Experimental): Administration of SNK01 4ⅹ10^9 cells/dose 8 times at an interval of 1 week + Administration of Cytotoxic Chemotherapy (GC) up to 4 cycles at an interval of 3 weeks
  Interventions: Biological: SNK01 (Super Natural Killer Cells 01); Drug: GC
- SNK01 (4ⅹ10^9 cells) + GC + Cetuximab (Experimental): Administration of SNK01 4ⅹ10^9 cells/dose 8 times at an interval of 1 week + Administration of Cytotoxic Chemotherapy (GC) up to 4 cycles at an interval of 3 weeks + Weekly administration of Cetuximab until the disease progresses or unacceptable toxicity develops
  Interventions: Biological: SNK01 (Super Natural Killer Cells 01); Drug: GC; Biological: Cetuximab
- SNK01 (6ⅹ10^9 cells) + GC (Experimental): Administration of SNK01 6ⅹ10^9 cells/dose 8 times at an interval of 1 week + Administration of Cytotoxic Chemotherapy (GC) up to 4 cycles at an interval of 3 weeks
  Interventions: Biological: SNK01 (Super Natural Killer Cells 01); Drug: GC
- SNK01 (6ⅹ10^9 cells) + GC + Cetuximab (Experimental): Administration of SNK01 6ⅹ10^9 cells/dose 8 times at an interval of 1 week + Administration of Cytotoxic Chemotherapy (GC) up to 4 cycles at an interval of 3 weeks + Weekly administration of Cetuximab until the disease progresses or unacceptable toxicity develops
  Interventions: Biological: SNK01 (Super Natural Killer Cells 01); Drug: GC; Biological: Cetuximab

INTERVENTIONS:
Biological: SNK01 (Super Natural Killer Cells 01) — Investigational Product : SNK01 (Super Natural Killer Cells 01) Principal Component : Autologous Natural Killer Cell To induce anti-tumor immunity in Locally advanced or Metastatic Non-small Cell Lung Cancer Patients who have failed prior TKI therapy for EGFR, ALK, or ROS1 Gene Mutation and to strengthen the Antibody-Dependent Cellular Cytotoxicity (ADCC) of Cetuximab, 4x10^9 or 6x10^9 cells are infused through the veins of the subjects within 45 minutes (±15 minutes) per 100 mL total 8 times at intervals of one week.
Drug: GC — Gemcitabine; 1000mg/m2, Day 1, Day 8, 4-cycle administration, Mixed with normal saline 50ml and administered into a vein for 30 min.
  Carboplatin; AUC 5, Day 1, 4-cycle administration, Mixed with 5% Dextrose 200ml and administered into a vein for 1 hour.
  Other Names: Cytotoxic Chemotherapy
Biological: Cetuximab — First administration: 400mg/m2 Subsequent administration: 250mg/m2 (Premedication before administration*) Weekly Administration continues until the disease progresses or unacceptable toxicity develops.
  400mg/m2: Administered into a vein for 120 minutes 250mg/m2: Administered into a vein for 60 minutes
  Arms: SNK01 (4ⅹ10^9 cells) + GC + Cetuximab; SNK01 (6ⅹ10^9 cells) + GC + Cetuximab

SUMMARY:
This clinical trial is a Single-Center, Open, Phase I/IIa Clinical Trial conducted to evaluate the safety and anti-tumor activity of SNK01 and GC +/- Cetuximab administered in combination to Locally advanced or Metastatic Non-small Cell Lung Cancer Patients who have failed prior Tyrosine Kinase Inhibitor (TKI) therapy at least once.

After the start of the clinical trial, the first 3 subjects complete the enrollment in Cohort 1 in serial order and then 3 subjects are enrolled in Cohort 2 in serial order. After this, Cohorts 1, 3 and Cohorts 2, 4 are independently processed and subjects are enrolled in serial order when new cohorts start and/or replacement subjects are required. For the subjects who are additionally enrolled after the DLT evaluation and the MTD is determined in each dose cohort, no DLT evaluation is conducted.

The subjects allotted to each cohort are administered with the SNK01 manufactured from peripheral blood mononuclear cells total 8 times over a period of about 10 weeks. Combined administration of SNK01 starts from the Cycle 2 (Week 4) of Cytotoxic Chemotherapy and SNK01 is administered at an interval of 1 week starting from the day after the administration of Cytotoxic Chemotherapy and/or Cetuximab (Visit 5-1, D23).

When no disease progression is confirmed at EOT (End of Treatment), disease progression is checked until the clinical trial is over. The adverse events which have occurred during the study period are monitored until the date when the investigator judges that no monitoring is required as the symptom has disappeared or there is no further change in the symptom or the 30th day (±3 d) from the latest date of the administration among Gemcitabine, Carboplatin and Cetuximab after the EOT, whichever comes first.

For all the subjects enrolled in the present clinical trial, safety is checked in accordance with CTCAE V5.0 and effectiveness is checked in accordance with RECIST V1.1 through the vital signs, laboratory test, adverse events, etc. during the study period.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically diagnosed with Locally advanced or Metastatic Non-small Cell Lung Cancer (TNM 8th edition). However, recurrent Non-small Cell Lung Cancer is also allowed.
* one or more gene mutations among EGFR, ALK, and ROS1
* TKI treated for EGFR, ALK, or ROS1 gene mutation at least once or whose progressive disease is confirmed during or after completion of the treatment
* platinum based chemotherapy (excluding Gemcitabine), other chemotherapy or immunotherapy besides TKI treatment before. (Those who have undergone neoadjuvant chemotherapy or adjuvant chemotherapy are also allowed.)
* remaining toxicity resulting from previous anti-cancer therapy is grade 1 or lower in accordance with CTCAE V5.0. However, those who suffer from alopecia not lower than grade 2 or neuropathy of grade 2 related to previous platinum based chemotherapy are allowed to be enrolled.
* voluntarily decided to participate in the present clinical trial and put their signature on a subject's consent form before start of the trial
* 20 years of age or older
* at least one lesion measurable by RECIST v1.1
* life expectancy is 3 months or longer
* Eastern Collaborative Oncology Group (ECOG) performance status is 0 or 1 when screened
* adequate blood and terminal organ functions
* For fertile women: Those who have agreed to maintain abstinence (refraining from sextual intercourses with men) or use a contraceptive measure of which the annual failure rate is lower than 1 % during the treatment period and for minimum 6 months (180 days) after the last administration of SNK01, GC, or Cetuximab. Women who have had their first menstrual period, not yet reached a post-menopausal state (amenorrhea for longer than 12 months in succession without cause other than menopause) and have not undergone surgical sterilization (ovariectomy or hysterectomy) and under the age of 55 with follicle stimulating hormone (FSH) levels of less than 40 mIU/mL are considered as fertile women. However, women who have already confirmed menopause are excluded. The examples of the contraceptive measures of which the failure rate is lower than 1 % include the following: Bilateral Tubal Ligatio, male sterilization, established and appropriate use of hormonal contraception that inhibits ovulation, hormone releasing IUD (IntraUterine Device) and copper IUD. The reliability of abstinence should be evaluated based on the clinical trial period and the daily life-style preferred by the patient. Periodic abstinence (example: calendar method, ovulation, and post-ovulation body temperature measurement method) and coitus interrupts are not acceptable contraceptive measures.
* For men: Those who have agreed to maintain abstinence (refraining from sextual intercourses with women) as defined below, use contractiptive measures, and abstain from sperm donation. Men with a fertile spouse should maintain abstinence or use of condoms and additional contraceptive measures during the treatment period and for minimum 4 months (120 days) after the last administration of SNK01, GC or Cetuximab so that the annual failure rate is lower than 1 %. Men should abstain from sperm donation during this period. The reliability of sexual abstinence should be evaluated based on the study period and the normal life-style preferred by the patient. Periodic abstinence (example: calendar method, ovulation, and post-ovulation body temperature measurement method) and coitus interrupts are not acceptable contraceptive measures.
* adapt themselves to the Protocol according to the judgment of the investigator

Exclusion Criteria: Subjects who fulfill ANY of the following criteria will not be enrolled into the study:

* have taken a drug for another clinical trial or participated in another clinical trial within 30 days prior to the enrollment
* have taken Cetuximab to cure Non-Small Cell Lung Cancer
* a systemic or partial antineoplastic therapy is scheduled during the period of the present study
* previous treatments meet the following criteria:

  1. Those who have undergone systemic Cytotoxic Chemotherapy, administration of a biologic agent, or a surgery within 3 weeks prior to the enrollment date
  2. Those who have undergone Breast Radiotherapy of which the radiation exceeds 30 gray (Gy) for treatment of Non-small Cell Lung Cancer within 6 months prior to the enrollment date
  3. Those who have undergone Palliative Radiotherapy on the regions to which a lung cancer is metastasized (bone, brain, etc.) within 1 week before the enrollment date
  4. Those who have undergone therapy of EGFR TKIs (Gefitinib, Erlotinib, Afatinib, Osimertinib, etc.), ALK TKIs (Crizotinib, Ceretinib, Alectinib, Brigatinib, etc.) and/or ROS1 TKIs (Crizotinib, etc.) within 2 weeks of the enrollment date
* an anamnesis of a known allergic reaction or a serious allergic reaction to Gemcitabine, Carboplatin, or another platinum containing compound, Cetuximab or a monoclonal antibody
* uncured or active Central Nervous System (CNS) metastasis confirmed by screening and previous CT or MRI evaluation. However, the patients who have cured or symptomless CNS metastasis are allowed to be enrolled if they meet all the following criteria:

  1. if a lesion exists on the region other than the area of CNS metastasis that can be evaluated or measured by RECIST V1.1;
  2. if it is radiologically confirmed before the enrollment that the lesion is stabilized after the area of CNS metastasis has been treated;
  3. if the patients have no anamnesis of intracranial hemorrhage or myelorrhagia; and
  4. if the patients have clinically stable symptomless lesion for minimum 2 weeks after treatment of the CNS metastasis and stopping use of anticonvulsant or steroid.
* an active autoimmune disorder within 2 years prior to the enrollment date which requires systemic treatment
* undergone allogeneic stem cell or solid-organ transplant before
* an interstitial lung disease or pneumonitis which requires orally or intravenously administered steroid treatment
* have been inoculated or plan to be inoculated with live attenuated influenza vaccine within 30 days prior to the enrollment date
* an active infection that requires systemic treatment through intravenous administration
* positive for HIV, HBV, or HCV
* a medical history related to psychiatry or an anamnesis of drug abuse or alcoholism that will affect participation in the present clinical trial
* an anamnesis of another malignant tumor within recent 5 years. However, patients with a non-melanoma skin carcinoma appropriately treated or with another cancer that shows no evidence of the disease after receiving potential treatment and for which no evidence of recurrence is found for 5 years from the starting point of the treatment by the doctor in charge are allowed to be enrolled.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-07-08 (Actual); Primary Completion 2023-05-26 (Estimated); Study Completion 2023-05-26 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of the dose of SNK01 + GC + (or Cetuximab) | 28 days
  Dose-Limiting Toxicity assessment
Adverse event | Up to 12 months
  Adverse event (AE)

SECONDARY OUTCOMES:
Progression-free survival | every 12 weeks, up to the time of death or tumor progression, maximum 24 months
  Progression-Free Survival (PFS)
Disease Control Rate | every 12 weeks, up to the time of death or tumor progression, maximum 24 months
  Disease Control Rate (DCR)
objective response rate | every 12 weeks, up to the time of death or tumor progression, maximum 24 months
  objective response rate (ORR)
Time to progression | every 12 weeks, up to the time of death or tumor progression, maximum 24 months
  Time to progression (TTP)
Duration of response | every 12 weeks, up to the time of death or tumor progression, maximum 24 months
  Duration of response (DoR)
QoL | every 12 weeks, up to the time of death or tumor progression, maximum 24 months
  EoRTC QLQ-C30
QoL | every 12 weeks, up to the time of death or tumor progression, maximum 24 months
  EORTC QLQ-LC13

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi MG, Son GW, Choi MY, Jung JS, Rho JK, Ji W, Yoon BG, Jo JM, Kim YM, Ko DH, Lee JC, Choi CM. Safety and efficacy of SNK01 (autologous natural killer cells) in combination with cytotoxic chemotherapy and/or cetuximab after failure of prior tyrosine kinase inhibitor in non-small cell lung cancer: non-clinical mouse model and phase I/IIa clinical study. J Immunother Cancer. 2024 Mar 27;12(3):e008585. doi: 10.1136/jitc-2023-008585. PMID 38538093